CLINICAL TRIAL: NCT02537132
Title: "New Perspectives of Adaptation to Non-Invasive Ventilation (NIV) in Amyotrophic Lateral Sclerosis (ALS)"
Brief Title: "New Perspectives of Adaptation to NIV in ALS"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Fondazione Salvatore Maugeri (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDG_ALS1H_01
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Non Invasive Ventilation (NIV); Amyotrophic Lateral sclerosis (ALS); adaptation; home care
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Acclimatization

ARMS (2):
- Home Group (Experimental): Adaptation and training to Non Invasive Ventilation (NIV) (not less than five sessions), at home
  Interventions: Other: Adaptation and training to Non Invasive Ventilation (NIV)
- Outpatient Group (Active Comparator): Adaptation and training to Non Invasive Ventilation (NIV) (not less than five sessions), at the outpatient clinic
  Interventions: Other: Adaptation and training to Non Invasive Ventilation (NIV)

INTERVENTIONS:
Other: Adaptation and training to Non Invasive Ventilation (NIV) — Each person recruited after a respiratory evaluation (baseline spirometry and supine, maximal inspiratory and expiratory pressures (MIP / MEP) or sniff nasal inspiratory pressure (SNIP), 6 Minute Walking Test (6MWT) -if still ambulatory, arterial blood gas, nocturnal polygraphy) will be adapted to Non Invasive Ventilation (NIV). Moreover, the subject will be brought to the management of bronchial secretions (under the terms set out herein) during not less than five outpatient or house accesses, depending on who is randomly assigned to the experimental group or the control group. These accesses will take place weekly, for a period of two months, considering both the needs and the patient's clinical condition.

SUMMARY:
The purpose of this study is to demonstrate that the adaptation to the Non Invasive Ventilation (NIV) at home is not worse when compared with an adaptation performed in inpatient settings.

ELIGIBILITY:
Inclusion Criteria:

* ALS diagnosis according to the criteria of El Escorial;
* Clinical indication to NIV (nocturnal hypoventilation and respiratory muscle weakness confirmed according to the criteria normally accepted);
* No respiratory infection within 3 months
* Severe disability (ALS-FRS <31);
* Age > 18 years;
* The voluntary participation to the Study.

Exclusion Criteria:

-- Previous episodes of pneumothorax;

* Comorbid cardiac and / or renal important
* Severe cognitive impairment;
* Refusal of the patient at the time of Informed Consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2018-01

PRIMARY OUTCOMES:
Change from baseline in adherence NIV in ALS patients at baseline, 2 and 4 months as measured by monthly means and standard deviations of hours of use of Non Invasive Ventilation (NIV) | Baseline + after 2 and 4 months from the recruitment
  The primary outcome the time of adherence to NIV defined as actual use of NIV for not less than 150 hours / month.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Michele Vitacca, Lumezzane, Brescia
  - Paolo Banfi, Milan